CLINICAL TRIAL: NCT00866554
Title: Phase II Study of Bicalutamide and Dutasteride for Prostate Cytoreduction Prior to Permanent Implant I-125 Prostate Brachytherapy
Brief Title: Efficacy and Toxicity of Bicalutamide and Dutasteride vs. Standard Care for Prostate Cytoreduction for Brachytherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, André-Guy Martin, MD MSC FRCP(C) Radio-oncologue, Curiethérapeute Professeur Associé, Université Laval, CHU de Quebec-Universite Laval
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DUT112661; Health Canada-112661 (Other Grant/Funding Number: GSK)
Record Dates: First submitted 2009-03-19; First posted 2009-03-20 (Estimated); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Prostate Cancer; Erectile Dysfunction; Lower Urinary Tract Symptoms
Keywords: Prostate; Brachytherapy; Cytoreduction; Sexual function; Toxicity
MeSH Terms: conditions — Prostatic Neoplasms; Erectile Dysfunction; Lower Urinary Tract Symptoms | interventions — bicalutamide; Dutasteride; Tamoxifen

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- LHRH agonist (Active Comparator): Administration of a 3-month treatment with an LHRH agonist (chosen by the treating radiation oncologist) and Bicalutamide 50 mg daily for the first month of treatment with the LHRH agonist.
  Interventions: Drug: administration of a LHRH agonist and Bicalutamide
- Dutasteride, Bicalutamide, Tamoxifen (Experimental): Administration of Dutasteride given at dose of 0.5 mg daily starting three months prior to day of implant procedure and continued for 3 months up until procedure.
  Bicalutamide: given at a dose of 50 mg daily for 3 the same 3 month period as dutasteride
  Tamoxifen: given at dose of 10 mg daily for 3 months that dutasteride and bicalutamide are administered.
  Interventions: Drug: administration of Bicalutamide, Dutasteride and Tamoxifen

INTERVENTIONS:
Drug: administration of a LHRH agonist and Bicalutamide — 3-month treatment with an LHRH agonist chosen by the treating radiation oncologist and Bicalutamide 50 mg daily for the first month of treatment with the LHRH agonist.
  Other Names: Bicalutamide(Casodex)
  Arms: LHRH agonist
Drug: administration of Bicalutamide, Dutasteride and Tamoxifen — Dutasteride given at dose of 0.5 mg daily starting three months prior to day of implant procedure and continued for 3 months up until procedure.
  Bicalutamide: given at a dose of 50 mg daily for 3 the same 3 month period as dutasteride
  Tamoxifen: given at dose of 10 mg daily for 3 months that dutasteride and bicalutamide are administered.
  Other Names: Bicalutamide (Casodex); Dutasteride (Avodart); Tamoxifen (Nolvadex)
  Arms: Dutasteride, Bicalutamide, Tamoxifen

SUMMARY:
The purpose of this study is to determine if a combination of neoadjuvant dutasteride and bicalutamide has the same efficacy and less toxicity than standard treatment with an LHRH agonist and bicalutamide for prostate cytoreduction prior to permanent implant brachytherapy.

DETAILED DESCRIPTION:
Permanent implant prostate brachytherapy is recognized as the treatment method for prostate cancer that results in the least amount of sexual side effects including erectile dysfunction (ED). However prostate brachytherapy is often limited to patients with a prostate volume less than 50cc because of dosimetric and technical considerations. To counter this fact patients with a prostate larger than 50cc are offered neoadjuvant hormonal therapy to reduce their prostate volume to a value less than 50cc. The pharmacological method most often employed involves treatment with an LHRH agonist, which also involves multiple adverse effects for patients including ED in the majority of patients.

This approach may also involve other disadvantages including a possibility of increased cardiovascular mortality a possible increase in urinary toxicity and a reduction in health-related quality of life in patients treated with neoadjuvant hormonal therapy. Despite theses facts, neoadjuvant hormonal therapy remains essentially the sole method used to reduce prostate volume prior to prostate brachytherapy. One study has evaluated the efficacy of a neoadjuvant regimen without an LHRH agonist, comprised of Dutasteride and Bicalutamide to reduce prostate volume. This treatment could theoretically have fewer effects on sexual function and quality of life and could also possibly reduce urinary toxicity of brachytherapy. Nonetheless, these factors have never been evaluated. The cytoreductive efficacy of Bicalutamide and Dutasteride have never been directly compared to standard treatments. The current study is necessary to determine the effects of a neoadjuvant regimen of Bicalutamide and Dutasteride on prostate volume, sexual function, urinary toxicity and quality of life as compared to standard treatment. If it can be determined that there is an advantage with Bicalutamide and Dutasteride this regimen could become a standard of care for prostate cytoreduction prior to brachytherapy.

ELIGIBILITY:
Inclusion Criteria:

* Male sex
* Diagnosis of prostate adenocarcinoma as confirmed by prostate biopsy
* Prostate cancer with stage T1a, T1b T2a or T2b Nx Mx as determined by clinical examination
* Gleason score of 6 or less or 7 (3+4)*

  * If Gleason score is 7(3+4) patient must have less than 30% of biopsied tissue positive
* Serum PSA of ≤ 15ng/ml during the month before study entry
* Prostate volume ≥ 45cc
* Normal serum testosterone during the month before study entry
* Availability for treatment and follow-up visits
* Having signed required consent form before study entry

Exclusion Criteria:

* Abnormal Liver Function tests (>2x normal AST or ALT and/or >1.5x normal bilirubin)
* Prostate volume less than 50 cc
* History of hormonal treatment including any of the above: LHRH agonists, antiandrogens during the year before study entry
* Use of a 5 alpha reductase inhibitor for more than one month during the year prior to study entry
* History of pelvic irradiation
* History of past chemotherapy
* History of TURP
* History of past treatment for prostate cancer
* Known hypersensitivity to Dutasteride or Bicalutamide
* Co-morbid disease possibly compromising treatment compliance
* History of DVT or pulmonary embolism
* Anticoagulation with coumarin
* Inability to give consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-03; Primary Completion 2019-03 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Total prostate volume | 3 months after start of therapy
  Trans rectal ultra sound 3 dimensional volume evaluation

SECONDARY OUTCOMES:
EPIC questionnaire urinary function and bother scores | baseline, pre-implant, 6 weeks post-implant, 3,6,12,18 and 24 months post-implant
  Expanded Prostate Cancer Index Composite
EPIC questionnaire sexual function and bother scores | baseline, pre-implant, 6 weeks post-implant, 3,6,12,18 and 24 months post-implant
  Expanded Prostate Cancer Index Composite
EPIC questionnaire bowel function and bother scores | baseline, pre-implant, 6 weeks post-implant, 3,6,12,18 and 24 months post-implant
  Expanded Prostate Cancer Index Composite
EPIC questionnaire hormonal function and bother scores | baseline, pre-implant, 6 weeks post-implant, 3,6,12,18 and 24 months post-implant
  Expanded Prostate Cancer Index Composite
IPSS scores | baseline, pre-implant, 6 weeks post-implant, 3,6,12,18 and 24 months post-implant
  International Prostate Symptom Score (I-PSS)
Acute urinary retention rates | 0 to 6 months post-implant
  Common Terminology Criteria for Adverse Events (CTCAE)
SF-12 Quality of life questionnaire results | baseline, pre-implant, 6 weeks post-implant, 3,6,12,18 and 24 months post-implant
  International Quality of Life Assessment - Short Form
Rate of gynecomastia and breast tenderness | 6 weeks pre-implant, pre-implant, 6 weeks post-implant, 3,6,12,18 and 24 months post-implant
  Common Terminology Criteria for Adverse Events (CTCAE)
Serum testosterone | 3 months pre-implant, pre-implant, 3,6,12,18 and 24 months post-implant
  testosterone blood level
Anemia | baseline, pre-implant, 3,6,12,18 and 24 months post-implant
  haemoglobin blood level
Abnormal liver function tests | 6 weeks pre-implant, pre-implant, 3 months post-implant
  Blood level of Alanine transaminase (ALT), Aspartate transaminase (AST), Alkaline phosphatase (ALP), Bilirubin, Gamma-glutamyltransferase (GGT), L-lactate dehydrogenase (LD).
Serum PSA | baseline, pre-implant, 3,6,12,18 and 24 months post-implant
  serum testosterone blood level
Adverse events recording | 6 weeks pre-implant, pre-implant, 6 weeks post-implant, 3,6,12,18 and 24 months post-implant
  Common Terminology Criteria for Adverse Events (CTCAE)

CONTACTS AND LOCATIONS:
Overall Officials: Andre-Guy Martin, MD, Principal Investigator — CHUQ-Hotel-Dieu de Québec
Locations (1):
- CHUQ- Hotel-Dieu de Quebec, Québec, Quebec, Canada